CLINICAL TRIAL: NCT06368050
Title: Implementation of an Evidence-Based Intervention to Improve Head Impact Safety in Youth Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Childress Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00067187.2
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-04

CONDITIONS: Head Injury; Sport Injury
Keywords: Sport Safety; Youth Football; Head Impact Exposure
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Unexposed practice group
- Experimental - practice structure intervention (Experimental): Athletes of teams at the 12U and 13U level pilot testing the intervention program. On-field activity will be monitored with head impact sensors and video to evaluate the effectiveness of the intervention program.
  Interventions: Behavioral: practice structure intervention

INTERVENTIONS:
Behavioral: practice structure intervention — practice structure intervention
  Arms: Experimental - practice structure intervention

SUMMARY:
The objective of this study is to evaluate the feasibility of implementing an evidence-based intervention program, COmmunities Aligned to reduce Concussion and Head impact exposure (COACH) on a larger scale. Coaches of 12U (12 years old and under), and 13U (13 years old and under) teams within six youth football organizations will pilot test the intervention. Aim 1 will conduct focus groups with coaches, parents, and organizational leaders to assess organizational needs, capacity, and readiness to adopt the intervention program. Aim 2 will evaluate the effectiveness of the intervention program at reducing HIE and injuries and evaluate implementation success. Aim 2 results (intervention outcomes) are reported herein.

DETAILED DESCRIPTION:
Coaches of teams at the 12U and 13U levels within the six youth football organizations will be invited to pilot test the intervention program. Intervention outcomes will be compared to historic controls (K25HD101686 - NCT04908930). Video taken at all practices will be used to monitor team activities of 12U and 13U teams across all organizations participating in the intervention; incidence of injuries will be monitored across all teams. Athletes (n=30) enrolled across two of six participating teams will be recruited to participate in parallel biomechanical and video data collection to evaluate the frequency and severity of head impacts experienced throughout the season. Biomechanical data will be collected using instrumented mouth guards and verified with video. Preliminary effectiveness will be measured by the percentage of coaches who choose to adopt and maintain the intervention program. Head impact exposure and injury rates will be compared across the intervention and control teams.

ELIGIBILITY:
Inclusion Criteria:

* All athletes participating on the prospective teams will be eligible for the study, including those with braces longer than 6 months

Exclusion Criteria:

* Athletes will be excluded from participation if they have had braces less than 6 months, or have dental appliances that may impede the fit of the mouthpiece device (e.g., Herbst Appliance).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Number of practice head impacts | Month 3
  Number of verified direct head impacts measured in practice over the entire season.
Number of practice head acceleration events | Month 3
  Number of verified direct and indirect head acceleration events measured in practice over the entire season.
Practice head impact rate | Month 3
  Rate of verified direct head impacts per athlete per practice
Practice head acceleration even rate | Month 3
  Rate of verified direct and indirect head acceleration events per athlete per practice
Median linear acceleration | Month 3
  Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of median linear acceleration.
Median rotational acceleration | Month 3
  Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of median rotational acceleration.
Median rotational velocity | Month 3
  Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of median rotational velocity
95th percentile linear acceleration | Month 3
  Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of 95th percentile linear acceleration
95th percentile rotational acceleration | Month 3
  Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of 95th percentile rotational acceleration
95th percentile rotational velocity | Month 3
  Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of 95th percentile rotational velocity

SECONDARY OUTCOMES:
Feasibility of Intervention Measure (FIM) Values | up to 13 weeks
  Perceived feasibility - higher values denote better feasibility - total range 0 - 5
Acceptability of Intervention Measure (AIM) Values | up to 13 weeks
  Higher values denote better acceptability - total range 0 - 5
Number of practices the intervention was implemented as prescribed | up to 13 weeks
  The extent to which the intervention was implemented as prescribed. Descriptive data and inferential statistics will be used. Common themes will be grouped, and qualitative data indexed and charted
Average minutes per practice of live time | up to 13 weeks
  Minutes per practice spent on live tackling

CONTACTS AND LOCATIONS:
Overall Officials: Jill Urban, PhD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT06368050/ICF_000.pdf